CLINICAL TRIAL: NCT06586723
Title: Impact Trial of Helping Educational Leaders Mobilize Evidence
Acronym: HELM 2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Responsible Party: Principal Investigator, Jill Locke, Associate Professor: School of Medicine, Psychiatry, University of Washington
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Health Services Research
Other Study IDs: STUDY00020559
Record Dates: First submitted 2024-08-27; First posted 2024-09-19 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2024-09

CONDITIONS: Child Development; Child Behavior
MeSH Terms: conditions — Child Behavior

STUDY DESIGN:
Intervention Model Description: All schools that participate in the study will receive PBIS. Additionally, half of the schools will be randomized to receive HELM, an additional implementation support intervention.
Who Masked: Outcomes Assessor
Masking Description: PBIS coaches will be masked to HELM randomization
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- PBIS (Active Comparator): Positive Behavioral Interventions and Supports (PBIS) is an evidence-based, multi-tiered, problem-solving, and team-based framework designed to build a continuum of supports to promote all students' social emotional behavioral health.
  Interventions: Behavioral: PBIS
- HELM (Experimental): Helping Educational Leaders Mobilize Evidence (HELM) is an implementation strategy for promoting building-level implementation leadership, implementation climate, and high-fidelity delivery of evidence-based practices
  Interventions: Behavioral: PBIS; Other: HELM

INTERVENTIONS:
Behavioral: PBIS — Positive Behavioral Interventions and Supports (PBIS) is an evidence-based, multi-tiered, problem-solving, and team-based framework designed to build a continuum of supports to promote all students' social emotional behavioral health.
Other: HELM — Helping Educational Leaders Mobilize Evidence (HELM) is an implementation strategy for promoting building-level implementation leadership, implementation climate, and high-fidelity delivery of evidence-based practices
  Arms: HELM

SUMMARY:
Social, emotional, and behavioral (SEB) problems occur frequently among elementary school students, dramatically impede student outcomes, and have been exacerbated by the COVID-19 pandemic. Evidence based practices exist to address student SEB needs, prevent problems, and ensure academic success. However, the implementation of these programs in schools is frequently incomplete, uneven, and occurs with insufficient fidelity to ensure positive effects for students due to significant implementation barriers across multiple levels. The purpose of this Impact Trial is to test the effectiveness of the Helping Educational Leaders Mobilize Evidence (HELM) implementation strategy in school-wide implementation of a Tier 1 evidence-based practice (EBP) - Positive Behavioral Interventions and Supports (PBIS).

ELIGIBILITY:
Inclusion Criteria:

* School Districts: School districts in Washington State committed to implementing PBIS in its elementary schools
* Educators: Educators working in a public elementary school within an enrolled school district.

Exclusion Criteria:

* Schools with previous HELM exposure will be excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2028-08-31 (Estimated); Study Completion 2028-08-31 (Estimated)

PRIMARY OUTCOMES:
PBIS Fidelity (Tiered Fidelity Inventory) | Baseline, 9 months, 12 months
  The Tiered Fidelity Inventory (TFI) is a 45-item tool used to provide a valid, reliable, and efficient measure of the extent to which school personnel are applying the core features of PBIS. The TFI is a group-assessment completed by a schoolwide system planning team with external facilitation with strong internal consistency. The scoring criteria for each individual item ranges from 0-3 (0=Not Implemented, 1=Partially Implemented, 3=Fully Implemented); higher scores indicate better outcome.

SECONDARY OUTCOMES:
Implementation Leadership: School Implementation Leadership Scale (SILS) | Baseline, 9 months, 12 months
  The SILS has 24 items loading onto 8 subscales: Proactive, Knowledgeable, Supportive, Perseverant, Communication, Vision, Available, and Distributed Leadership. The scoring criteria for each individual item ranges from 0-4; higher scores indicate better outcome.
Implementation Climate: School Implementation Climate Scale (SICS) | Baseline, 9 months, 12 months
  The SICS includes 21 items loading onto 7 subscales: Focus on EBP, Educational Support for EBP, Recognition for EBP, Rewards for EBP, Use of Data to Support EBP, Existing Supports for EBP, and EBP Integration. The scoring criteria for each individual item ranges from 0-4; higher scores indicate better outcome.
Implementation Cost | Baseline, 9 months, 12 months
  This survey asks educators how much time they spent on study-related procedures each week. Inputs will include time, supplies, travel, overhead, and costs associated with HELM training/coaching meetings, including pre-work, scheduling, and attending meetings; as well as costs associated with PBIS training and delivery.
Academic Engagement, Prosocial Behavior, and Problem Behavior: Modified Direct Behavior Rating (DBR) | Baseline, 9 months, 12 months
  The DBR will be used in which teachers observe and rate their classroom's overall academic engagement (i.e., actively or passively participating in the classroom activity, 0-100%), disruptive behavior (i.e., interrupting activities, 0-100%), and prosocial behavior (i.e., following directions, 0-100%; Chafouleas et al., 2012).
Student Academic Outcomes | Baseline, 9 months, 12 months
  Standardized academic test scores will be derived from administrative records.
Student Disciplinary Incidents | Baseline, 9 months, 12 months
  Number of office discipline referrals, suspensions, and expulsions will be derived from administrative records.
Student Attendance Rates | Baseline, 9 months, 12 months
  Student attendance rates will be derived from administrative records.
HELM Fidelity | Baseline, 9 months, 12 months
  As a manipulation check to document HELM intervention delivery, we will assess HELM fidelity using the HELM fidelity checklist (based on observations of recorded HELM trainings). HELM coaches will complete a standardized measure of dates specific steps were completed. Schools that achieve 80% or higher of the maximum possible score on all HELM fidelity criteria will be considered having received a full dose of HELM training and coaching.

CONTACTS AND LOCATIONS:
Overall Officials: Jill Locke, PhD, Principal Investigator — University of Washington; Aaron Lyon, PhD, Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Locke J, Williams NJ, Sridhar A, Ehrhart MG, Dopp A, Thirion M, Espeland C, Riddle B, Schmitz K, Hatch K, Buehler L, Lyon AR. Study protocol for testing the efficacy of the Helping Educational Leaders Mobilize Evidence (HELM) implementation strategy in elementary schools: a hybrid type 3 effectiveness-implementation randomized controlled trial. Implement Sci. 2025 Apr 24;20(1):17. doi: 10.1186/s13012-025-01429-4. PMID 40275358